CLINICAL TRIAL: NCT06308263
Title: Phase 1 Study to Evaluate the Mass Balance, Pharmacokinetics, Metabolism, Excretion and Absolute Bioavailability of Tuvusertib (M1774) Containing Microtracer 14C Tuvusertib in Participants With Advanced Solid Tumors (DDRIVER Solid Tumors 303)
Brief Title: Tuvusertib (M1774) Human Mass Balance and Absolute Bioavailability Study (DDRIVER Solid Tumors 303)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS201924_0003; 2022-502940-10-00 (Other: EU trial number)
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
Keywords: Ataxia telangiectasia mutated and Rad3-related (ATR) inhibitor; ADME; Tuvusertib (M1774)
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Period 1: Mass Balance: Tuvusertib + [14C]Tuvusertib microtracer (Experimental)
  Interventions: Drug: Tuvusertib [14C]Tuvusertib microtracer; Drug: Tuvusertib
- Period 1a: Absolute Bioavailability: Tuvusertib + [14C]Tuvusertib microdose bolus injection (Experimental)
  Interventions: Drug: Tuvusertib; Drug: Tuvusertib + [14C]Tuvusertib microdose bolus injection
- Period 2: Tuvusertib (Experimental)
  Interventions: Drug: Tuvusertib

INTERVENTIONS:
Drug: Tuvusertib [14C]Tuvusertib microtracer — Participants will receive single oral dose of Tuvusertib containing a [14C] Tuvusertib microtracer solution on Day 1 of period 1 under fasted conditions.
  Other Names: M1774
  Arms: Period 1: Mass Balance: Tuvusertib + [14C]Tuvusertib microtracer
Drug: Tuvusertib — Participants will also receive a single oral dose of Tuvusertib on Day 1 of Period 1 or Period 1a, and daily single oral dose of Tuvusertib for 2 weeks in 21 days cycle of Period 2.
  Other Names: M1774
Drug: Tuvusertib + [14C]Tuvusertib microdose bolus injection — In Period 1a, participants will receive on Day 1 of Period 1 a single oral dose of tuvusertib and an intravenous (IV) (14C) tuvusertib microdose as bolus injection.
  Other Names: M1774
  Arms: Period 1a: Absolute Bioavailability: Tuvusertib + [14C]Tuvusertib microdose bolus injection

SUMMARY:
This is a single sequence 2-period open label study in participants with advanced solid tumors. The purpose of Period 1 of this study is to assess the mass balance to determine drug-related entities present in circulation and excreta and provide a comprehensive understanding of biotransformation pathways and clearance mechanisms in participants with advanced solid tumors. The purpose of Period 1a is to assess the extent of ABA of tuvusertib and the mass balance, PK, metabolism, and elimination of 14C-tuvusertib after iv dosing in participants with advanced solid tumors. After either Period 1 or Period 1a; participants may enter an optional extension phase (Period 2) where participants will receive tuvusertib until disease progression or other criteria for study intervention discontinuation are met.

ELIGIBILITY:
Inclusion Criteria:

* Are histologically proven advanced solid tumors that are considered appropriate for treatment in Period 2 of this study, for which no effective standard therapy exists, or standard therapy has failed or cannot be tolerated
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) less than or equal to 1 (<=) 1
* Have evaluable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at Screening
* Are capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Uncontrolled or poorly controlled arterial hypertension, symptomatic congestive heart failure (New York Heart Association Classification more than equal to (>=) Class III), uncontrolled cardiac arrhythmia, calculated Corrected QT interval (QTc) average using the QT Interval Corrected Using Fridericia's Formula (QTcF) more than (>) 480 msec; unstable angina pectoris, myocardial infarction, or a coronary revascularization procedure, cerebral vascular accident, transient ischemic attack, or any other significant vascular disease within 180 days of study intervention start
* Presence of toxicities due to prior anticancer therapies (e.g. radiotherapy, chemotherapy, immunotherapies, Et cetera (etc.)) that do not recover to (<=) Grade 1 with the exception of toxicities that do not pose a safety risk to the participant in the judgment of the Investigator (e.g. ongoing Grade 2 alopecia)
* Treatment with live or live attenuated vaccine within 30 days of dosing (non-replicating vector vaccines are permitted)
* Participation in a study involving administration of 14C-labeled compound(s) within last 6 months prior to start of study intervention
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Period 1: Percent Urinary Recovery (feurine) Of Total Radioactivity (TRA) Over the Entire Period Of Collection | Pre-dose up to 312-336 hours post dose
Period 1: Percent Fecal Recovery (fefeces) Of TRA Over the Entire Period Of Collection | Pre-dose up to 312-336 hours post-dose
Period 1: Percent Total Recovery in Urine and Feces (fetotal) Of TRA Over the Entire Period of Collection | Pre-dose up to 312-336 hours post-dose
Period 1 and 1a: Maximum Observed Plasma Concentration (Cmax) Of Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1 and 1a: Time to Reach Maximum Plasma Concentration (Tmax) Of Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1 and 1a: Area Under the Plasma Concentration-Time Curve from Time Zero to the Time of the Last Quantifiable Concentration (AUC0-tlast) Of Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1 and 1a: Area Under the Plasma Concentration-Time Curve (AUC) from Time Zero Extrapolated to Infinity (AUC0-inf) Of Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1 and 1a: Apparent Terminal Half-Life (t1/2) Of Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1 and 1a: Apparent Total Body Clearance (CL/F) Of Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1 and 1a: Apparent Volume of Distribution (Vz/F) Of Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1: Maximum Observed Concentration (Cmax) of TRA in Plasma and Whole Blood | Pre-dose up to 336 hours post-dose
Period 1: Time to Reach Maximum Concentration (tmax) of TRA in Plasma and Whole blood | Pre-dose up to 336 hours post-dose
Period 1: Area Under Concentration-Time Curve from Time Zero to the Time of the Last Quantifiable Concentration (AUC0-tlast) of TRA in Plasma and Whole Blood | Pre-dose up to 336 hours post-dose
Period 1: Area Under the Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUC0-inf) of TRA in Plasma and Whole Blood | Pre-dose up to 336 hours post-dose
Period 1: Apparent Terminal Half-Life (t1/2) of TRA in Plasma and Whole Blood | Pre-dose up to 336 hours post-dose
Period 1a: Ratio of Dose Normalized AUC0-infinity of Tuvusertib and 14C Tuvusertib in Plasma | Pre-dose up to 336 hours post-dose
Period 1a: Initial Concentration (C0) at Time Zero After Bolus Intervention Administration of 14[C] Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1a: Maximum Observed Concentration (Cmax) at Intravenous Administration of 14 [C] Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1a: Total Body Clearance (CL) Following at Intravenous Administration of 14[C] Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1a: Volume of Distribution (Vz) during the terminal phase following intravenous administration of 14[C] Tuvusertib | Pre-dose upto 336 hours post-dose
Period 1a: Volume of Distribution at Steady State (Vss) Following at Intravenous Administration of 14[C] Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1a: Area Under the Plasma Concentration-Time Curve from Time Zero to the Time of the Last Quantifiable Concentration (AUC0-tlast) at Intravenous Administration of 14[C] Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1a: Area Under the Plasma Concentration-Time Curve (AUC) from Time Zero Extrapolated to Infinity (AUC0-inf) at Intravenous Administration of 14[C] Tuvusertib | Pre-dose up to 336 hours post-dose
Period 1a: Apparent Terminal Half-Life (t1/2) at Intravenous Administration of 14[C] Tuvusertib | Pre-dose up to 336 hours post-dose

SECONDARY OUTCOMES:
Period 1,1a,2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Treatment-Related AEs, Abnormal Laboratory Parameters, abnormal Vital Signs and abnormal 12-Lead Electrocardiogram (ECG) Findings | Baseline up to safety follow up (assessed up to approximately 21 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Pharmaceutical Research Associates Magyarország Kutatás - Fejlesztési Kft., Klinikai Farmakológiai Vizsgálóhely, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research.
  Further information on how to request data can be found on our website bit.ly/IPD21.

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?idMS201924_0003
- See also: US Medical Information website, Medical Resources — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html